CLINICAL TRIAL: NCT01637766
Title: Selective Intra-arterial Chemotherapy in the Treatment Strategy of Metastatic Spinal Disease
Brief Title: Intra-arterial Chemotherapy for Spinal Metastases
Acronym: SIAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0807009906
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Spinal Diseases; Spinal Metastases; Spinal Tumors
Keywords: Spinal Metastases; Spinal Metastatic Disease; Cord Compression; Intra-arterial Chemotherapy; Spinal Tumors
MeSH Terms: conditions — Spinal Diseases; Spinal Cord Neoplasms; Spinal Cord Compression | interventions — Melphalan; Infusions, Intra-Arterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Selective intra-arterial chemotherapy (Experimental): Subjects recruited to this study will receive intra-arterial injections of chemotherapy (melphalan) in the branches of the arteries feeding the metastatic spinal tumor. Subjects will receive general anesthesia or conscious sedation. A catheter will be guided using X-ray from the femoral artery at the top of the leg to the arteries of the spine. A dye will be injected through the catheter to show the arteries in greater detail. The chemotherapy is then injected into the tumor. We will inject the maximum systemic dose adjusted to white blood count and platelet count. Subjects will undergo three cycles of chemotherapy three to six weeks apart.
  Interventions: Drug: Melphalan (intra-arterial infusion)

INTERVENTIONS:
Drug: Melphalan (intra-arterial infusion) — Patients will undergo a minimally invasive procedure called spinal angiography. This procedure will identify the arteries feeding the tumor causing cord compression and will determine whether chemotherapy can be safely infused.
  The chemotherapy will be infused via a tiny soft plastic tube (called "microcatheter") at the tumor site over approximately 30 minutes.
  The drug of choice is melphalan (trade name Alkeran) at a maximum dose of 16mg/m2, adjusted for white cell count, platelet count and renal function.
  We will perform up to three intra-arterial chemotherapy treatments in 3-6 week intervals, based on the results of complete blood counts.
  Other Names: Alkeran

SUMMARY:
Metastatic malignant tumors comprise the vast majority of spinal tumors in adults. The most devastating complication of spinal metastatic disease (SMD) is invasion of the spinal canal and compression of the spinal cord or the nerve roots of the cauda equina, resulting in a clinical entity known as cord compression that manifests with progressive loss of motor function and sensation in the legs, as well as bladder and bowel incontinence.

The treatment of spinal metastases is mostly palliative with the goals of improving or maintaining neurologic function, achieving local tumor control, and spinal stability. Most patients with spinal metastatic disease are currently treated effectively with radiation therapy and/or surgery with good results. There are however certain limitations in the current treatment of SMD. Radiation therapy has two important limitations: 1) if the targeted SMD is in close proximity the spinal cord, delivery of high radiation doses is contraindicated as it may cause radiation-induced damage to the spinal cord (myelopathy, and 2) there is limit on the cumulative amount of radiation dose, which means that recurrent tumors may not be amenable to repeat radiation therapy. As far spinal surgery is concerned, the main limitation is that some patients are not fit for surgery because of medical co-morbidities.

This phase I clinical research trial will test the hypothesis that a new minimally invasive treatment called spinal intra-arterial chemotherapy (SIAC) can be safely applied in patients with SMD.

DETAILED DESCRIPTION:
To date, there is no effective systemic therapy for spinal metastases, and the goal of treatment is to achieve local control of the tumor. Despite advances in radiation therapy, there is still a subgroup of patients that cannot be effectively treated with radiation because of close proximity of the tumor to the spinal cord. In addition, in cases of recurrent tumors, some patients cannot be re-treated because they reached the maximum allowed radiation dose. Surgery is the alternative treatment for these patients, but some tumors do recur after surgery while some patients have comorbidities that make surgery a high-risk procedure.

Based on our prior experience with selective IA chemotherapy for the treatment of ocular retinoblastoma and the high local control rates achieved with selective IA injection of chemotherapy in recurrent limb melanoma (limb infusion and limb perfusion) we expect that spinal intra-arterial chemotherapy with selective injection of Melphalan in the arteries feeding the metastatic disease is feasible and safe and may prove beneficial in achieving local control of the spinal tumor, preventing neurological compromise from cord compression. This minimally invasive approach can be used in patients in whom radiation therapy and surgery are contra-indicated and essentially have no other treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic diseases to the spine causing cord compression grades 1, and 2 who are not candidates for the standard treatment of radiation therapy or surgery.
* Patients older than 18 years old.
* Patients able to give informed consent.

Exclusion Criteria:

* MRI findings of grade 3 epidural cord compression.
* Rapidly worsening neurological symptoms.
* The vascular supply to the spinal cord (anterior and/or posterior spinal arteries) originates from the same segmental arteries (intercostal or lumbar arteries) supplying the tumor.
* Life expectancy less than 3 months.
* Pregnant or lactating patients.
* Female patients with inadequate contraception.
* History of severe allergy to contrast media.
* Renal insufficiency (Creatinine >1.5mg/dL)
* WBC < 3000 cells/ mm3
* Platelets < 75000 cells/ mm3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in whom intra-arterial chemotherapy is performed without severe complication. | 30 days

SECONDARY OUTCOMES:
Change in spinal epidural tumor size as depicted on the MRI scans after treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Athos Patsalides, Principal Investigator — Weill Cornell
Locations (1):
- Weill Cornell Medical College Department of Neurological Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No